CLINICAL TRIAL: NCT00591695
Title: Prospective, Randomised European Multicentric Study, Comparing Enteral Stent Followed by Elective Surgery Versus Emergency Surgical Treatment in Malignant Colonic Obstruction
Brief Title: Enteral Stents for Colonic Obstruction
Acronym: ESCO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: European Association for Endoscopic Surgery (Other)
Responsible Party: Principal Investigator, Alberto Arezzo, Assistant Professor of Surgery, European Association for Endoscopic Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAES-1
Record Dates: First submitted 2007-12-29; First posted 2008-01-11 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Malignant Colorectal Obstruction
Keywords: Malignant Colorectal Obstruction; Stent Bridge to Surgery
MeSH Terms: interventions — Elective Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): positioning in emergency of a prosthetic metallic self-expanding stent followed, in case of successful colic decompression, by an elective surgical (laparoscopic or open) resection of the tumour
  Interventions: Procedure: Stent bridge to surgery + elective surgery
- B (Active Comparator): emergency surgery performed in these ways: Resection followed by enterostomy (Hartmann procedure), 'On table' washing and primary anastomoses, Subtotal colectomy
  Interventions: Procedure: Emergency Surgery

INTERVENTIONS:
Procedure: Stent bridge to surgery + elective surgery — positioning in emergency of a metallic self-expanding stent followed, in case of successful colic decompression, by an elective surgical (laparoscopic or open) resection of the tumour
  Other Names: Colorectal stenting with metallic self-expanding stent + elective surgery
  Arms: A
Procedure: Emergency Surgery — Emergency surgery performed in these ways: Resection followed by enterostomy (Hartmann procedure), 'On table' washing and primary anastomoses, Subtotal colectomy
  Other Names: Resection followed by enterostomy (Hartmann procedure); 'On table' washing and primary anastomoses; Subtotal colectomy
  Arms: B

SUMMARY:
The purpose of this study is to verify whether stent positioning for malignant obstruction of the colon and rectum followed by elective surgery allows reduction of postoperative complications and hospital stay without worsening of evolution of the neoplastic illness, compared to emergency surgery.

Primary endpoint will be 60 days postoperative morbidity. Others endpoints will be postoperative mortality, length of hospital stay, need for analgesia.

DETAILED DESCRIPTION:
Introduction & background In emergency surgery, although surgical and resuscitation techniques were improved, the postoperative complications and mortality rates are still high and however higher than for those patients that underwent to elective surgery (1-3). Using a Metallic prosthesis stent in an obstructed colon allows to transform an emergency surgical case into an elective surgery case. This allows to restore the bowel transit and to operate in elective condition reducing morbidity, mortality and the need of an enterostomy (4-10).

Although there are recent outcomes on literature about use of a decompressive stent before surgery in obstructed patients from malignant colic tumours, there are no prospective and randomised studies were stent positioning followed by elective surgery is compared with emergency surgery.

Study design Prospective, randomized multicentric clinical trial where samples are patients with emergency room diagnosis of obstructing colonic neoplasm.

Once informed and obtained consent, patients will be included in the study and randomized in one of the two branches of the study: A.- enteral stent positioning followed by second time resection in the same hospital stay. B.- emergency surgical treatment consisting in Hartmann operation or resection with same time anastomosis. Results from transit reconstruction in patients underwent Hartmann operation will be considered in the study.

Short term clinical evolution control in order to determine postoperative morbility and mortality, hospital stay.

Follow-up will be performed to evaluate survival rate and disease free survival.

Endpoints To evaluate and compare the results obtained using enteral stent followed by elective surgery versus common emergency surgical techniques.

Primary endpoint will be 60 days postoperative morbidity. Others endpoints will be: postoperative mortality, length of hospital stay, need for analgesia. Long term follow up with specific instrumental controls (CT scan, US, colonoscopy or RX clysma) to identify disease recurrences or metastases as cost analysis and patient's quality of life will also be evaluated.

Statistics & randomization In prospective series analysed in different centres, the incidence of postoperative complications in patients underwent to emergency colonic surgery was 35%. The positioning of the stent associated to second time surgical elective treatment is characterized by 15% of morbidity (stent: 5%, surgery: 10%). The number of patients needed to carry on the study making statistically significant this difference (35% vs 15%) with an error alpha = 0.05 and beta = 0.2 and estimating a loss of 5% of the samples, is 72 patients in each group.

Randomization will be stratified for local extension of tumour (T4 vs others) and for presence or not of liver metastases.

Main selection criteria Inclusion of patients with malignant colonic obstruction localized between promontorium and splenic flexure and diagnosed by CTScan. Those patients with peritonitis, pneumoperitoneum, synchronic colonic tumour, pregnant or haemodynamic instability will be excluded.

Follow-up Same follow-up as patients diagnosed and treated for Colon Cancer following the protocol of each center, never less than 3 years. During follow-up required complementary studies will be performed in each case in order to evaluate local recurrence or distant metastases. Also quality of life and costs will be evaluated.

Expected results: reduction of postoperative complications and hospital stay in patients submitted to stent positioning without worsening of evolution of the neoplastic illness.

ELIGIBILITY:
Inclusion Criteria:

* malignant colonic obstruction localized between splenic flexure and 15 cm from anal margin diagnosed by CTScan.
* Possibility of endoscopy and stent location during next 24 h after diagnostic.
* Clinical occlusion to gas and faeces.
* Informed consent obtained from the patient or from a relative in case of inability.

Exclusion Criteria:

* Bowel perforation diagnosed by clinical exploration and complementary studies.
* Associated pathologies contraindicating general anaesthesia and/or haemodynamic instability.
* Impossibility to gain a valid informed consent or refusal from the patient.
* Patients with multiple liver metastases diagnosed by CTScan at the moment of diagnostic and not considered operable with curative intention following the standards of every center.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative complications | 60 days

SECONDARY OUTCOMES:
postoperative mortality | 30 days
success percentage of stent positioning in emergency | at stent positioning
percentage of complications related to stent positioning | at stent positioning
length of hospital stay | 3 months
quality of life and survival | 3 years
cost differences | 3 months
oncological results (local and distant recurrence rate) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mario Morino, Professor of Surgery, Principal Investigator — University of TORINO - European Association for Endoscopic Surgery; Eduardo M Targarona, Professor of Surgery, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (2):
- Department of Surgery, Minimally Invasive Surgery Center, University of Torino, Torino, Italy
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Derived] Arezzo A, Forcignano E, Bonino MA, Balague C, Targarona E, Borghi F, Giraudo G, Ghezzo L, Passera R, Morino M; collaborative ESCO study group. Long-term Oncologic Results After Stenting as a Bridge to Surgery Versus Emergency Surgery for Malignant Left-sided Colonic Obstruction: A Multicenter Randomized Controlled Trial (ESCO Trial). Ann Surg. 2020 Nov;272(5):703-708. doi: 10.1097/SLA.0000000000004324. PMID 32833762